CLINICAL TRIAL: NCT03121183
Title: Medico-economic Evaluation of Strategies for the Lead Extraction of Implantable Defibrillator and Pacemakers: a Retrospective Observational Study
Brief Title: Medico-economic Evaluation of Strategies for the Lead Extraction of Implantable Defibrillator and Pacemakers
Acronym: GAINE LASER
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-318
Record Dates: First submitted 2017-04-14; First posted 2017-04-20 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-04

CONDITIONS: Prosthesis-Related Infections; Equipment Failure; Heart Failure; Arrhythmias; Thrombosis
Keywords: Cardiology; Device Removal; Pacemaker; Defibrillators; Catheterization; Laser Therapy; Cost-Benefit Analysis
MeSH Terms: conditions — Prosthesis-Related Infections; Heart Failure; Arrhythmias, Cardiac; Thrombosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who have undergone an extraction of implantable pace
  Interventions: Device: Laser sheath; Behavioral: Implantable Cardiac Device lead extraction

INTERVENTIONS:
Device: Laser sheath — Patients who have undergone an extraction of implantable pacemaker or defibrillator leads whatever the indication for the period march 2015-2017
Behavioral: Implantable Cardiac Device lead extraction — Patients who have undergone an extraction of implantable pacemaker or defibrillator leads whatever the indication for the period march 2015-2017

SUMMARY:
The growing use and the expanding indications for cardiovascular implantable electronic devices (CIEDs) have been associated to an increase of device removal. The indications of CIEDs removal are infectious (55%) or noninfectious (45%) such as upgrading of devices, nonfunctional devices and thrombosis. Removal can be performed according to transvenous or surgical procedures. Transvenous lead removal (TLR) must be done by experimented cardiologists and respecting current consensus. TLR can be done with conventional techniques involving inserting locking stylets and telescoping sheaths around the pacing leads to separate them from the surrounding scar tissue. These conventional procedures have a success rate of ≈65%. TLR thanks to laser sheath has been validated and improved the success rate until >95%. However, the TLR from chronically implanted CIEDs still carries a significant risk of procedural failure, morbidity, and mortality, related to tearing of the great vessels and cardiac structures, even when performed by experienced operators. Even if the transvenous extraction using laser sheath seems to be more effective, this strategy would be more expensive.

Considering the availability of several strategies for TLR and the cost heterogeneity of procedures, a cost assessment in real life of these therapeutic strategies is essential for an optimal choice of therapeutic strategies.

DETAILED DESCRIPTION:
The study will compare the strategies of percutaneous extraction to surgical extraction.

* Mechanical percutaneous extraction is the conventional technique using locking stylets and telescoping sheaths around the pacing leads to separate them from the surrounding scar tissue.
* Laser-assisted lead extraction is most often used in complex procedures and dissolves rather than tear the scar tissue.
* Sternotomy is the surgical procedure used when leads cannot be removed by percutaneous extraction. It is rarely employed.

ELIGIBILITY:
Inclusion Criteria:

* - Patients who have undergone an extraction of implantable pacemaker or defibrillator leads whatever the indication for the period march 2013-2017

Exclusion Criteria:

* - None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Patients who have undergone an extraction of implantable pacemaker or defibrillator leads whatever the indication for the period march 2013-2017
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2018-04 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Direct medical cost | at day 1
  Overall cost of care according to the hospital perspective: drug treatment, medical device, catheterization lab occupancy, operating room occupancy, medical and nursing staff time, hospitalization

SECONDARY OUTCOMES:
Investment cost for the hospital and damping | at day 1
  annual projections: medical device and supplies
Type of intervention | at day 1
  mechanical percutaneous extraction, laser percutaneous extraction, surgical extraction
Indication of the intervention | at day 1
  infectious, technical failure or other
Extracted leads characteristics | at day 1
  number, type, age, failure
Patient characteristics | at day 1
  age, sex, origin (general hospital, university hospital, other)
Number and type of complications | at day 1
  tamponade, vascular rupture, haemothorax, equipment breakage, death…
percutaneous extraction | at day 1
  number of surgical transformation (sternotomy)
Duration of hospitalization | at day 1
  pre and post-extraction
Duration of extraction procedure and fluoroscopy | at day 1
  for percutaneous extraction
quotation ranking of each patient for revenue valuation | at day 1
  quotation ranking of each patient for revenue valuation
Number of rehospitalization | at day 1
  duration, cause and service

CONTACTS AND LOCATIONS:
Overall Officials: David BALAYSSAC, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France